CLINICAL TRIAL: NCT00852839
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Arm Study of 552-02 in Subjects With Dry Mouth Associated With Sjogren's Syndrome
Brief Title: A Safety and Efficacy Study of 552-02 in Subjects With Dry Mouth Associated With Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 552-207S
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2014-07

CONDITIONS: Dry Mouth Associated With Sjogren's Syndrome; Xerostomia
Keywords: Dry mouth; Sjogren's syndrome; Xerostomia
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 552-02 (Experimental)
  Interventions: Drug: 552-02
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to match oromucosal formulation of 552-02
  Arms: Placebo
Drug: 552-02 — The oromucosal formulation of 552-02 contains 552-02 (25 μg/mL), surfactant, flavoring agents, a humectant, and preservatives.
  Arms: 552-02

SUMMARY:
This clinical study is to determine whether daily administration of a formulation of 552-02 improves the dry mouth condition in subjects with primary Sjögren's syndrome.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to determine whether daily administration of an oromucosal formulation of 552-02 improves the global assessment of dry mouth, as assessed by visual analog scale (VAS), in subjects with primary Sjögren's syndrome.

The secondary objectives of this study are as follows:

* To evaluate the safety of daily administration of an oromucosal formulation of 552-02 in subjects with primary Sjögren's syndrome.
* To evaluate whether administration of an oromucosal formulation of 552-02 improves the subjective measurement of 6 different salivary functions, as measured using VAS, in subjects with primary Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80 years (inclusive), and capable of providing their written informed consent.
* Male subjects must be either not sexually active, surgically sterilized, or agree to use an appropriate "double-barrier" method during study participation and for at least 30 days after the completion of dosing.
* Non-pregnant female subjects must be either not sexually active, post-menopausal, surgically sterilized; or agree to use an appropriate "double-barrier" method; or are currently using a prescribed transdermal, injection, implant, or oral contraceptive for at least 30 days before study participation and at least 30 days after the completion of dosing.
* Good health, as determined by a medical history, a physical examination, a detailed oral examination, 12-lead ECG, and measurement of clinical chemistry, hematology, urinalysis, and serology data.
* Demonstrated minimal level of unstimulated whole mouth salivary flow (greater than or equal to 0.05 milliliters [ie, 0.05 grams] per 5 minutes).
* Demonstrated clinically significant, moderate to severe level of dry mouth at screening as determined by his/her score on a 100-mm global VAS of dry mouth symptoms with anchors ranging from 'not dry at all' (0) to 'dry as a desert' (100) as follows:
* Minimal VAS score of 50 mm at Visit 1.
* Diagnosis of primary Sjögren's syndrome.

Exclusion Criteria:

* Currently using a potassium-sparing diuretic antihypertensive drug that contains amiloride; spironolactone (e.g.,Aldactone, Novo-Spiroton, Spiractin, Spirtone, Verospiron or Berlactone); triamterene (e.g., Dyrenium); or plerenone (e.g., Inspra). Chronic use antihistamines will be permitted if started at least 30 days before Visit 1, and a stable dose is maintained throughout the trial.
* Started using systemic cholinergic secretagogues or tricyclic antidepressant drugs within 12 weeks before screening, is not on a stable dosing regimen for at least 14 days prior to the Screening visit, or who is unable to maintain stable dosing throughout the study.
* Unable to withhold the use of oral comfort agents (eg, Oasis, MouthKote, etc) following enrollment in the study (Visit 1).
* Shows evidence of a significant active or ongoing oral infection or other oral conditions (eg, lichen planus) that, in the opinion of the Investigator, might affect the safety of the subject or be exacerbated during study participation.
* Acutely infected salivary glands or suspected closure of the salivary glands.
* A condition that may confound the diagnosis of primary Sjögren's syndrome.
* Received an investigational drug within the past 30 days.
* Received 552-02 in a previous study.
* History of multiple drug allergies or allergy to any medicine chemically related to the study drug (eg, amiloride, Moduretic, Midamor, triamterene).
* Any clinically significant allergic disease, including food allergies, with the exception of nonactive hayfever.
* Present history of any clinically significant and uncontrolled neurologic, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, or hematological disorder or disease, or any other major disorder or disease, in the opinion of the Investigator.
* Sitting blood pressure at screening higher than 150/90 mmHg or lower than 100/50 mmHg after resting for 5 minutes.
* Sitting pulse rate at screening outside the range of 50 - 90 beats per minute (bpm) after resting for 5 minutes.
* Consumes more than 2 alcoholic drinks per day or has a significant history of alcoholism or drug/chemical abuse within the past 12 months.
* History of using tobacco products within the last 3 months.
* Has viral hepatitis or tests positively for the hepatitis B surface antigen (HBsAg) or hepatitis C (non-A, non-B) antibody, or a positive result for human immunodeficiency virus (HIV) antibodies.
* Positive serum pregnancy test or is nursing (female subjects only).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Global assessment of dry mouth, as assessed by visual analog scale (VAS), in subjects with primary Sjögren's syndrome. | 49 Days

SECONDARY OUTCOMES:
To evaluate the safety of daily administration of an oromucosal formulation of 552-02 in subjects with primary Sjögren's syndrome. | 49 Days

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - New England Research Associates, LLC, Trumbull, Connecticut
  - University of Florida College of Dentristy, Gainesville, Florida
  - Indiana School of Dentristy, Indianapolis, Indiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Winthrop University Hospital, Mineola, New York
  - AAIR Research Center, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oklahoma University, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Penn Rheumatology Associates, Philadelphia, Pennsylvania
  - Rheumatology Consultants, Knoxville, Tennessee
  - Arthritis Centers of Texas, Dallas, Texas
  - Univ. of Texas Health Science Center, San Antonio, Texas
  - Arthritis Northwest, Spokane, Washington